CLINICAL TRIAL: NCT07060846
Title: Endoscopic Versus Open Lumbar Discectomy in Diabetic Patients: A Randomized Controlled Trial
Brief Title: Endoscopic Versus Open Lumbar Discectomy in Diabetic Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Awad Mohamed Hegab, Lecturer of Neurosurgery, Faculty of Medicine, Al-Azhar University, Damietta, Egypt., Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DFM-IRB 00012367-25-06-009
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Endoscope; Open; Lumbar Discectomy; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): Patients will undergo endoscopic lumbar discectomy.
  Interventions: Procedure: Endoscopic lumbar discectomy
- Group II (Active Comparator): Patients will undergo an open lumbar discectomy.
  Interventions: Procedure: Open lumbar discectomy

INTERVENTIONS:
Procedure: Endoscopic lumbar discectomy — Patients will undergo endoscopic lumbar discectomy.
  Arms: Group I
Procedure: Open lumbar discectomy — Patients will undergo an open lumbar discectomy.
  Arms: Group II

SUMMARY:
This study aims to compare the endoscopic versus open lumbar discectomy in diabetic patients.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is a highly prevalent disease with the capacity to adversely affect nearly every major organ system. DM has been demonstrated as a risk factor for a variety of complications within medical and surgical spheres Open lumbar discectomy is the most common surgical discectomy technique and is considered by many to be the gold standard.

Endoscopic lumbar discectomy allowed spinal surgeons to decompress a symptomatic lumbar nerve root by using an endoscopic minimally invasive surgical approach.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 75 years.
* Both sexes.
* Patients suffering from prolapsed lumbar disc postero-lateral, single level disc herniation at L4-5 or L5-S1 level with low back pain and unilateral radiculopathy and failure of conservative treatment for 12 weeks

Exclusion Criteria:

* Extraforaminal disc herniation.
* Recurrent and/or multiple level discs prolapses.
* Spondylolisthesis.
* Prior lumbar surgery at the same spinal level.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-19 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Degree of low back pain | 48 hours postoperatively
  The patients will be evaluated clinically using Visual Analogue Score (VAS) for low back pain and radicular pain. VAS (0 represents "no pain" while 10 represents "the worst pain imaginable"). VAS will be assessed at 0, 4, 8, 12, 18, 24, 36 and 48 h postoperatively.

SECONDARY OUTCOMES:
Degree of radicular pain | 48 hours postoperatively
  The patients will be evaluated clinically using Visual Analogue Score (VAS) for radicular pain and radicular pain. VAS (0 represents "no pain" while 10 represents "the worst pain imaginable"). VAS will be assessed at 0, 4, 8, 12, 18, 24, 36 and 48 h postoperatively.
Length of hospital stay | 1 week postoperatively
  Length of hospital stay will be recorded from admission till discharge from hospital.
Intraoperative blood loss | Intraoperatively
  Intraoperative blood loss will be recorded.
Operative time | Intraoperatively
  Operative time will be recorded from the start of surgery till the end of surgery.
Wound length | Intraoperatively
  Wound length will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar University (Damietta), Damietta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: The data will be available upon a reasonable request from the corresponding author.
Access Criteria: After the end of study for one year.